CLINICAL TRIAL: NCT04327063
Title: A Double-blind Randomized Trial of Interpectoral Nerve Block (Pecs 1 and 2) With Ropivacaine Versus Placebo Before Breast Cancer Surgery: Effects on Acute Postoperative Pain. (MIRs 04)
Brief Title: MIRs 04 : Interpectoral Nerve Block With Ropivacaine Versus Placebo Before Breast Cancer Surgery
Acronym: MIRs 04
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IC 2019-04
Record Dates: First submitted 2020-03-09; First posted 2020-03-30 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Malignant Neoplasm of Breast
Keywords: Surgery conservative; Nerve block
MeSH Terms: conditions — Breast Neoplasms | interventions — Sodium Chloride; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Saline (30 mL maximum)
  Interventions: Drug: Saline
- Ropivacaïne (Experimental): Ropivacaïne 5 mg/mL (not to exceed 3 mg/kg and 30 ml of maximal volume)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Saline — Injection of the solution of Saline not exceeding 30 mL of maximal volume.
  Other Names: NA Cl 0.9%
  Arms: Placebo
Drug: Ropivacaine — Dilution of Ropivacaine 7.5 mg/ml to 5 mg/ml not to exceed 3 mg/kg of maximal dose and 30 ml of maximal volume
  Other Names: Naropeine
  Arms: Ropivacaïne

SUMMARY:
Compare the effect of ropivacaine versus placebo pectoral nerve block (Pecs 1 and 2) on acute pain after tumorectomy plus sentinel lymph node dissection on one day surgery.

DETAILED DESCRIPTION:
Before surgery, the 3rd interpectoral space will be identified. After aspiration, half of the solution of Ropivacaine 5 mg/ml not exceeding 3 mg/kg of maximal dose and 30 ml of maximal volume or saline (not exceeding 30 ml of maximal volume) will be injected into the interpectoral space underneath the pectoralis major muscle for the Pecs 1 block. The other half of the solution will be injected above the serratus anterior muscle at the third rib.

Evaluation of the percentage of patients treated with step 2 or 3 analgesics during the three postoperative hours.

ELIGIBILITY:
Inclusion Criteria:

1. Women with non-metastatic invasive breast carcinoma or breast carcinoma in situ treated by breast-conserving surgery (tumorectomy) with sentinel node technique on one day surgery.
2. Age between 18 and 85 years.
3. ASA class 1, 2 or 3
4. Signed informed consent form.

Exclusion Criteria:

1. Ongoing neoplasm or history of neoplasm other than breast cancer with the exception of: basal cell carcinoma, cervical carcinoma in situ, other treated cancer that has not relapsed during the 5 years preceding inclusion in the trial.
2. Axillary dissection planned during surgery planning
3. All bilateral surgery the day of Pecs administration
4. Metastatic breast carcinoma at diagnosis (M1).
5. Allergy to local anesthetics and morphine.
6. Use of analgesics during the 12 hours preceding the surgical procedure.
7. History of ipsilateral surgery during the previous 6 months.
8. History of substance abuse.
9. Pregnant woman or breastfeeding.
10. Subjects deprived of their liberty or under guardianship (including temporary guardianship).
11. Subjects no covered by social security scheme
12. Experiencing any psychiatric condition or major cognitive impairment that may hamper completion of self-reported questionnaires.

There is no prohibition for people to take part simultaneously in another search and there is no exclusion cause at the end of the research period

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
To compare the effect of ropivacaine versus placebo pectoral nerve block (Pecs 1 and 2) on acute pain after tumorectomy plus sentinel lymph node dissection on one day surgery | 3 hours
  Percentage of patients treated with step 2 or 3 analgesics during the first three postoperative hours after tumorectomy plus sentinel lymph node dissection, between the group with Ropivacaïne and the group with placebo

SECONDARY OUTCOMES:
Evaluation of acute pain at rest and after shoulder movement until 48 postoperative hours | 48 hours
  VAS Scale (0 to 10 : 0 = no pain and 10 = Worst pain possible) at rest and after shoulder movement every 30 minutes during the first three postoperative hours in the PACU and the day surgery unit and then at home every 6 hours for the first 48 postoperative hours .
Evaluation of acute pain until 48 postoperative hours | 48 hours
  Brief Pain Inventory Questionnaires at 48 hours will be collected with VAS Scale (0 to 10 : 0 = no pain and 10 = Worst pain possible)
Evaluation of patient's satisfaction on pain management | 48 hours
  Scale of satisfaction ( 0 to 10 : 0 = very bad and 10 = excellent) of the pain management at 48 post-operative hours
Evaluation of Remifentanil consumption during anesthesia | 3 hours
  Total dose of Remifentanil during anesthesia for a bispectral index between 40-60 or Analgesia Nociception Index (ANI) > 60%
Evaluation of analgesic consumption during the first 48 postoperative hours | 48 hours
  Consumption of Ketoprofene in systematic, Paracetamol if VAS>3 and Tramadol if analgesia is not enough during 48 postoperative hours
Evaluation of the incidence of nausea and vomiting during the first 48 postoperative hours | 48 hours
  Incidence of nausea and vomiting during the first 48 postoperative hours
Evaluation of complications of Pecs during 48 postoperative hours | 48 hours
  Complications of Pecs block: pneumothorax, nerve injury, hypotension, vascular puncture and systemic toxicity of local anaesthetic (seizures, etc.) collected
Evaluation of the incidence of serious adverse events during 30 days | 30 days
  Number of serious adverse events during 30 days after Pecs administration

CONTACTS AND LOCATIONS:
Overall Officials: Pierre FUMOLEAU, PhD, Study Director — Institut Curie
Locations (4):
- France (4):
  - Centre Jean Perrin, Clermont-Ferrand
  - Institut Curie, Paris
  - Hopital Tenon, Paris
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Result] Albi-Feldzer A, Gayraud G, Dureau S, Auge M, Lemoine A, Raft J. Efficiency of interpectoral and pectoserratus plane blocks for breast surgery: A randomized controlled trial. J Clin Anesth. 2025 Apr;103:111805. doi: 10.1016/j.jclinane.2025.111805. Epub 2025 Mar 10. PMID 40068583